CLINICAL TRIAL: NCT03636698
Title: Clinical Research: Effect of Chorioamnionitis on Platelet Activation and Placental Vessel Among Preterm Infants by Wnt-Flt1 Signal Pathway
Brief Title: Effect of Chorioamnionitis on Platelet Activation and Placental Vessel Among Preterm Infants by Wnt-Flt1 Signal Pathway
Status: Completed | Type: Observational
Sponsor: Guangdong Women and Children Hospital (Other)
Responsible Party: Principal Investigator, yangjie, Chief of Neontology Dept, Guangdong Women and Children Hospital
Other Study IDs: Guangdong W&C Hospital
Record Dates: First submitted 2018-08-01; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2016-06

CONDITIONS: Chorioamnionitis; Placenta Diseases; Thrombocytopenia; Preterm Infant
MeSH Terms: conditions — Chorioamnionitis; Placenta Diseases; Thrombocytopenia; Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — the placentas and cord blood after delivery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chorioamnionitis Group: preterm infants were born to mothers with chorioamnionitis
  Interventions: Other: chorioamnionitis
- Control Group: preterm infants were born to mothers without chorioamnionitis
  Interventions: Other: chorioamnionitis

INTERVENTIONS:
Other: chorioamnionitis — It is a observation research. We didn't intervene anything. The chorioamnionitis groups included the infants whose mothers were diagnosed chorioamnionitis by placental histopathology.

SUMMARY:
Objective:The purpose of this study was to explore the effect and mechanism of maternal chorioamnionitis on placental microvasculature and platelet activation among preterm infants by activating Wnt-Flt1 signal pathway .

Methods:With clinical randomized controlled trial (RCT), the cases were matched with 1:1 according to gestational age and divided into 2 groups according to the placental pathology result: chorioamnionitis group and control group. (1) To observe the platelet parameter, birth weight, thrombrocytopenia and hemorrhage complication, such as intracranial hemorrhage, retinal hemorrhage, pulmonary hemorrhage and gastrointestinal hemorrhage. (2) To observe the miscrovascular density (MVD) in placenta, platelet activating factor (CD62p,CD63) and thrombopotetin (TPO) in preterrn infants.The placental MVD was assessed by immunohistochemical method. The platelet activating factors were detected by flow cytometry. TPO was detected by ELISA. (3) To observe Wnt5a, Flt1 and VEGF in placenta and fetal circulation.The measurement data were analyzed by pair t test and conditional logistic regression. Pearson correlation analysis was used for relationship.

DETAILED DESCRIPTION:
The exclusive criteria included :(1) born to mother with no any other maternal complications; (2) no congenital abnormalities and neonatal asphyxia; (3) died or discharged within 72 hours.

ELIGIBILITY:
Inclusion Criteria:

1. gestational age<37weeks
2. admitted to the NICU at Guangdong Women and Children Hospital, with a date of birth from June 2016 to December 2016
3. whose mothers were diagnosed chorioamnionitis by placental histopathology

Exclusion Criteria:

1. born to mother with no any other maternal complications
2. no congenital abnormalities and neonatal asphyxia;
3. died or discharged within 72 hours.

Min Age: 1 Hour | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Chorioamnionitis contributes to the high morbidity and mortality in preterm infants, thrombocytopenia is one of the acute morbidity
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Placental Microvascular Density(%) | 24 hours
  Placental Microvascular Density (by placental histopathology)

SECONDARY OUTCOMES:
Incidence Hemorrhage Disease (%) | through study completion, an average of half year
  intraventricular hemorrhage (IVH), retinal hemorrhage, pulmonary hemorrhage and gastrointestinal hemorrhage
Wnt5a in Placenta(IOD) | 24 hours
  by placental histopathology
mean platelet volume(MPV) | 24 hours
  MPV (Fl)
platelet distribution width(PDW) | 24 hours
  PDW (%)
Platelet counts (PLT) | 24 hours
  PLT (10^9/L)
Thrombopoietin (cord blood) | 24 hours
  TPO(ng/ml)
Platelets Activation Factors in cord blood | 24 hours
  CD62p(%)
Flt1 in Placenta(IOD) | 24 hours
  by placental histopathology
VEGF in Placenta(IOD) | 24 hours
  by placental histopathology
Wnt5 in infants (ng/ml) | 24 hours
  test them by Elisa from cord blood
Flt1 in infants (ng/ml) | 24 hours
  test them by Elisa from cord blood
VEGF in infants (ng/ml) | 24 hours
  test them by Elisa from cord blood